CLINICAL TRIAL: NCT01003197
Title: Novel Preoperative Score Predicting Outcome Following Liver Resection
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Breitenstein Stefan, Dr. med., Department of Visceral- and Transplantation Surgery
Other Study IDs: StV 2009
Record Dates: First submitted 2009-10-27; First posted 2009-10-28 (Estimated); Last update posted 2009-10-28 (Estimated); Status verified 2009-10

CONDITIONS: Serious Complications Following Liver Resection
Keywords: Development; Validation; Prediction Score; Complication; Liver resection; develop and validate a score to predict serious complications following liver resection using pre-operative risk factors.

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- complication group < III
- complication group >= III

SUMMARY:
To develop and validate a score to predict serious complications following liver resection using pre-operative risk factors.

DETAILED DESCRIPTION:
Liver surgery is associated with a substantial rate of complications. Early identification of patients at risk of serious complications is important in order to adapt therapeutic strategies and to improve quality. The purpose of this study is to develop and validate a score to predict serious complications following liver resection using pre-operative risk factors.

ELIGIBILITY:
Inclusion Criteria:

* >= 18 years
* liver resection

Exclusion Criteria:

* Trauma cases

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HPB center Zurich, Switzerland
Sampling Method: Probability Sample
Dates: Start 2009-02; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
develop and validate a score to predict serious complications following liver resection using pre-operative risk factors. | postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Breitenstein, Dr. med., Principal Investigator — Department of Visceral and Transplantation Surgery, University Hospital of Zurich
Locations (1):
- Department of Visceral and Transplantation Surgery, University Hospital of Zurich, Zurich, Canton of Zurich, Switzerland